CLINICAL TRIAL: NCT06077942
Title: FX Shoulder Solutions Retrospective / Prospective Clinical Study
Status: Recruiting | Type: Observational
Sponsor: FX Shoulder Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: FXShoulder2022-01
Record Dates: First submitted 2023-09-26; First posted 2023-10-11 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Rotator Cuff Syndrome of Shoulder and Allied Disorders; Osteoarthritis Shoulder; Fracture, Shoulder
Keywords: Osteoarthritis; Roartator Cuff; Fracture; Arthroplasty
MeSH Terms: conditions — Shoulder Fractures; Osteoarthritis; Fractures, Bone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Subjects: Subjects implanted with the shoulder replacement medical devices manufactured by FX Shoulder Solutions and distributed by FX Shoulder Solutions.
  Interventions: Device: FX Artificial Shoulder Prosthesis

INTERVENTIONS:
Device: FX Artificial Shoulder Prosthesis — Humelock II Anatomic Shoulder System, Humelock II Reversible Shoulder System, Humelock Reverse Shoulder System, Humeris Shoulder System, Easytech Anatomical Shoulder System, PRCT II Fracture Plate, V-135

SUMMARY:
Subjects implanted with the shoulder replacement medical devices manufactured by FX Shoulder Solutions and distributed by FX Shoulder Solutions.

DETAILED DESCRIPTION:
To evaluate patient outcomes following shoulder replacement with FX Shoulder Solutions medical devices To demonstrate effectiveness, safety and survivorship of FX Shoulder Solutions medical devices To provide data and analysis to FX Shoulder Solutions to meet regulatory requirements.

To provide data and analysis for presentations, abstracts, publications and other public release of results.

Clinical data in the Investigator's clinic notes and patient files regarding demographics, baseline medical and shoulder status, surgical procedure and implant components, and any completed postoperative clinical data will be collected retrospectively as data for the Study following signed patient consent and enrollment into the study.

Each patient will be evaluated prospectively, and clinical data collected at the first baseline clinical evaluation using the protocol specified evaluations following study enrollment with successive postoperative evaluations in accordance with the postoperative intervals.

ELIGIBILITY:
Inclusion Criteria:

* Received an FX Shoulder Solutions replacement medical device in accordance with the Indications for Use based upon surgeons' determination and standard of care for the selected device system beginning January 1, 2018, through June 30, 2023.

Exclusion Criteria:

* Patient who does not meet the inclusion criteria above

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who received the study devices implanted by the Investigator in accordance with the Indications for Use beginning January 1, 2018, through June 30, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2032-12-30 (Estimated); Study Completion 2032-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who are at a minimum of 2 years postoperative follow-up based upon the following composite clinical success (CCS) of the Patient Reported Outcome Surveys and Investigator Range of Motion (ROM) assessments. | 10 years
  * Adjusted Constant Score > 70
  * No continuous radiolucency or device migration/subsidence
  * No revision surgery or removal
  * No serious device related adverse event
  The Study will continue to follow patients prospectively to 10 years postoperative to track survivorship.

SECONDARY OUTCOMES:
Adjusted Constant Score | 3, 6, 12, 24 months, 5 and 10 years.
  The Constant-Murley score (CMS) is a validated 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient. The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion (40 points) with the subject completing the assessment prior to the Investigator completing their part of the assessment. The higher the score, the higher the quality of the function.
  An Adjusted Constant score will be calculated using normalized values to account for age and gender, as based upon anatomical gender at birth.
QuickDASH | 3, 6, 12, 24 months, 5 and 10 years.
  QuickDASH measures an individual's ability to complete tasks, absorb forces, and severity of symptoms. The QuickDASH tool uses a 5-point Likert scale from which the patient can select an appropriate number corresponding to his/her severity level/ function level. The higher the score, the higher the function and lower pain in the patient.
American Shoulder and Elbow Surgeon (ASES) | 3, 6, 12, 24 months, 5 and 10 years.
  ASES is a validated patient-reported outcome which is composed of 10 functional questions and one pain VAS. The total score is of 100 maximum points and weighted evenly between pain and function
Visual Analog Scale (VAS). A validated measurement of pain in a patient where 0 indicates no pain and 100 indicates severe pain. The VAS is a straight horizontal line of fixed length. | 3, 6, 12, 24 months, 5 and 10 years
  A validated measurement of pain in a patient where 0 indicates no pain and 100 indicates severe pain. The VAS is a straight horizontal line of fixed length.
Range of Motion | 3, 6, 12, 24 months, 5 and 10 years.
  ROM - The patient performs active movements in all functional planes for the shoulder.
  Includes flexion, extension, abduction, adduction and internal and external rotation. Investigator estimates the range of movement and compares the affected with the unaffected shoulder and the normal expected range.
Number of Participants Who Have a Secondary Surgical Intervention (SSI) | 24 months and at 5 and 10 years
  SSI's are re-operations, revisions, and removals.
Device Related Adverse Events. | 24 months and at 5 and 10 years postoperative
  An adverse event that is related to the use of a device.
Serious Adverse Event | 24 months and at 5 and 10 years postoperative
  1. Led to a death,
  2. Resulted in life threatening illness or injury*
  3. Resulted in patient hospitalization or prolongation of existing hospitalization,
  4. Resulted in patient disability or permanent damage or required intervention to prevent permanent impairment/damage
  5. Led to a congenital abnormality or birth defect
Serious Adverse Device Effects (SADE) | 24 months and at 5 and 10 years postoperative.
  Adverse device effect that has resulted in any of the consequences characteristic of a serious adverse event.
Number of Participants with Radiographic Reviews and Assessments. | 24 months, at 5 years and 10 years postoperative
  Monitor implant integrity and signs of implant loosening

OTHER OUTCOMES:
Primary Effectiveness Endpoint | 24 months
  The primary safety endpoint is the occurrence of any serious, device-related adverse event through 24 months of follow-up defined as an onset date before or on 730 days following the index surgery. For the primary endpoint, device-related will be defined as definite, probable, or possible relationship to the device.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Rogers, BS, Study Director — FX Shoulder Solutions
Locations (2):
- United States (2):
  - OrthoArizona, Gilbert, Arizona
  - Advanced Orthopedics Institute, The Villages, Florida

IPD SHARING:
Plan to Share IPD: Undecided